CLINICAL TRIAL: NCT01328652
Title: A Randomized, Double-blind, Placebo-controlled Study of Dexlansoprazole to Treat Laryngopharyngeal Reflux and Lingual Tonsil Hypertrophy
Brief Title: Dexlansoprazole to Treat Laryngopharyngeal Reflux and Lingual Tonsil Hypertrophy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Advanced Center for Specialty Care (Other)
Collaborators: Takeda (Industry)
Responsible Party: Michael Friedman, MD, Head and Neck and Cosmetic Surgery, Inc.and Advanced Center for Specialty Care
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004 10/10
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Laryngopharyngeal Reflux; Hypertrophy of Lingual Tonsil
Keywords: LPR; LTH
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Dexlansoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Pump Inhibitor (Experimental): Treatment with dexlansoprazole 60 mg once daily for 3 months
  Interventions: Drug: dexlansoprazole

INTERVENTIONS:
Drug: dexlansoprazole — dexlansoprazole 60 mg once daily for 3 months
  Other Names: proton pump inhibitor; Dexilant

SUMMARY:
Main Hypothesis: The investigators hypothesize that measurements of lingual tonsil tissue (LTT) thickness will decrease following treatment with once daily oral dexlansoprazole 60 mg in patients diagnosed with laryngopharyngeal reflux (LPR) and lingual tonsil hypertrophy (LTH) compared to matched controls receiving placebo.

Primary endpoints include:

* 24-hour oropharyngeal pH testing, pre- and post-treatment
* Mean lingual tonsil tissue (LTT) thickness, pre- and post-treatment, as determined by CT scan of the base of tongue

Secondary endpoints include:

* Reflux Finding Score (RFS) on pre- and post-treatment endoscopy of the oropharynx
* Subjective outcome metrics for assessing LPR-related symptoms and associated quality of life
* Calgary Sleep Apnea Quality of Life Index
* Bed-partner assessment of snoring intensity according to a Visual Analog Scale
* Epworth Sleepiness Scale (ESS)
* Reflux Symptom Index (RSI)

Specific Aims: The primary objective of this study is to determine whether treatment of patients diagnosed with LPR and LTH with 3 months of PPI therapy reduces LTT thickness, as measured on CT scan of the tongue base.

The secondary objectives of this study are to:

* Evaluate changes in LPR-related symptoms and quality of life after therapy using the following subjective outcome metrics:

  * Calgary Sleep Apnea Quality of Life Index
  * Bed-partner assessment of snoring intensity according to a Visual Analog Scale
  * Epworth Sleepiness Scale
  * Reflux symptom index
* Correlate changes in LTT thickness with the following secondary endpoints:

  * Changes in the above subjective outcome metrics
  * Changes in endoscopic findings of LPR
  * Changes in 24-hour oropharyngeal pH study results

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE:

Detail: The backflow of gastric contents into the esophagus occurs in healthy people to a limited extent.[1] When the refluxed material transcends the upper esophageal sphincter and enters the laryngopharynx on a chronic basis, it is termed laryngopharyngeal reflux (LPR). LPR typically manifests as dysphonia, globus sensation, chronic cough, and throat irritation. Recent studies suggest that untreated LPR may be a cause of lingual tonsil hypertrophy (LTH), [2,3] which itself has been implicated as a contributing factor in obstructive sleep apnea-hypopnea syndrome (OSAHS).[4-6] Lingual tonsil tissue (LTT) is present to a variable degree in most individuals and tends to regress with age. Although standardized parameters for defining LTH have yet to be established, a recent study by Friedman et al [7] demonstrated that on average subjects with LPR, OSAHS, or both diseases had significantly thicker LTT on CT imaging than patients without either disease. Del Gaudio and coworkers [2] identified a trend between increasing severity of LTH and the frequency of reflux events, while Mamede et al [3] found a positive correlation between reflux symptoms and the degree of LTH.

LTH in the setting of LPR is thought to result from the edema and inflammation brought about by chronic exposure of the tissues to the refluxed acid. The resulting thickened and inflamed LTT may narrow the retrolingual airway, increasing the likelihood of airway obstruction and apneic events. Theoretically, increases in negative intrathoracic pressure secondary to the obstruction may, in turn, facilitate further LPR.

While the treatment of reflux has been shown to decrease indices of OSAHS severity in some patients, [8-10] a direct causal relationship between LPR and OSAHS has not been proven. Similarly, more evidence is necessary to elucidate the exact relationship between LPR and LTH. No study to date has investigated whether treatment of LPR reduces LTH. The investigators hypothesize that adequate treatment of LPR using a PPI in patients with LTH will result in a significant reduction in LTT thickness as well as improvement in OSAHS symptoms, if present. The proposed study is a randomized, double-blind, controlled trial to determine whether control of LPR reduces LTH and, as a corollary, improves OSAHS symptoms. Control of LPR will be determined by 24-hour oropharyngeal pH monitoring [11], and LTH will be measured on CT. While the length of time required for LTH regression to occur is not currently known, Reichel et al have found that 3 months of PPI therapy are typically necessary before improvement in LPR is seen. [12] Similarly, a study by Park et al showed a significantly greater rate of improvement or resolution of LPR symptoms when treatment with a PPI was for longer than 2 months. [13] PRELIMINARY STUDIES Preliminary Studies: In a previous study, the investigators utilized axial and sagittal CT images of the tongue base to measure LTT in patients with LPR, OSAHS, both conditions, or neither disease. The investigators found that patients with LPR, OSAHS, or LPR+OSAHS had significantly thicker LTT than patients without LPR or OSAHS. This study was presented at the 2009 Annual Meeting of the American Academy of Otolaryngology-Head and Neck Surgery and was published in the April 2010 issue of the journal Otolaryngology-Head and Neck Surgery.

RESEARCH DESIGN AND METHODS:

Overview: Prospective, randomized, double-blind, controlled study at a tertiary, university-affiliated medical center.

Sample size: In order to achieve a power of 0.95, a sample size of 40 subjects per group (80 total) was determined based on an a priori power analysis. The sample size stated in the original concept was an estimate and was not determined statistically.

Procedures: The study protocol begins after a patient has been diagnosed with laryngopharyngeal reflux (LPR) on the basis of routine history, physical exam, and diagnostic studies including 24-hour oropharyngeal pH monitoring with the Dx-pH Monitoring System (Restech, San Diego, California). Prospective candidates for the study will be asked to undergo CT imaging of the tongue base. Those who are subsequently diagnosed with lingual tonsil hypertrophy (LTH), as determined by mean lingual tonsil tissue (LTT) thickness greater than 3.0 mm on axial and sagittal views, will be eligible for enrollment, providing they meet the additional inclusion criteria listed above. The enrollment period is expected to last 12 months, and the total duration of the study is expected to be 18 months.

Once an eligible patient has agreed to participate in the study and provided informed consent, s/he will be randomly assigned to the experimental or control group according to a 1:1 ratio. Patients as well as the practitioner administering treatment will be blinded to patient group assignments. Patients in the experimental group will be started on a 3-month regimen of once daily oral dexlansoprazole 60 mg. Patients in the control group will receive a placebo once daily by mouth for the same length of time. Following completion of the 3-month treatment regimen, patients from both groups will undergo repeat 24-hour oropharyngeal pH testing and CT of the tongue base. Endoscopic findings of LPR will also be recorded before, monthly during treatment and after treatment using the Reflux Finding Score (RFS). A 3-month treatment period was chosen based on previous studies, which have shown failure of symptom resolution after shorter lengths of time. Once enrolled, patients will be seen in clinic approximately every four weeks. Treatment with cimetidine 200 mg PO BID will be offered as a rescue medication to patients of either group whose LPR symptoms worsen during the study. Once started, cimetidine, as well as study drug (dexlansoprazole or placebo) will be continued for the duration of the study. At study conclusion, all patients will be re-evaluated for continued treatment, based on the effectiveness of dexlansoprazole (after unblinding) and need for rescue medication (dexlansoprazole and placebo). If cimetidine fails to offer relief, the subject will be withdrawn from the study and other treatment options will be offered.

The Calgary Sleep Apnea Quality of Life Index (CSAQLI), visual analog scale for snoring (VAS), and Epworth Sleepiness Scale (ESS) will be used as subjective outcome metrics. These questionnaires are validated tools for assessing symptoms of obstructive sleep apnea/hypopnea syndrome (OSAHS) and associated quality of life. The Reflux Symptom Index (RSI), a validated instrument for assessing reflux symptoms, will also be administered along with the other questionnaires both prior to initiating therapy and again at the end of the 3-month period.

Data analysis and Interpretation:

Statistical analysis will focus on determining whether lingual tonsil tissue size differs before and after therapy. Mean lingual tonsil tissue size will be calculated along with standard deviation and student t test will be used to determine statistical significance.

Analysis will also examine the mean change in four subjective metrics, (1) Calgary Sleep Apnea Quality of Life Index, (2) Visual Analog Scale of snoring, (3) Epworth Sleepiness scale, and (4) Reflux Symptom Index. Again, means and standard deviations will be calculated and student t test will be used to assess statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LPR and LTH confirmed by 24-hour pharyngeal pH monitoring and CT of the tongue base, respectively
* Age > 20 and < 60 years
* Failure (in the opinion of the patient and treating physician) of current treatment regimen and willingness (by the patient) to discontinue all concurrent therapies for LPR whether prescription, over-the-counter, or herbal, and to remain off of these treatments for the entire course of the study

Exclusion Criteria:

* Pregnancy or anticipated pregnancy (confirmation of non-pregnant status will be made by urine human chorionic gonadotropin level)
* Lactation
* History or diagnosis of moderate to severe hepatic disease (based on liver function testing performed at screening adjusted for age, gender, race, concomitant medications and comorbidities
* Current or within the previous (12 mo) usage of a proton pump inhibitor
* Concurrent use of any medications, which interact adversely with dexlansoprazole or other proton pump inhibitors (e.g., penicillins, digoxin, iron salts, azole antifungals, atazanavir, tacrolimus, clopidogrel, etc.)
* Allergy or sensitivity to dexlansoprazole (or other proton pump inhibitor) or cimetidine (or other H2 blocker)
* History of laryngeal and/or pharyngeal surgery
* Preexisting voice or swallowing disorder not related to LPR
* Smoking
* Neoplastic or infectious processes that are systemic or localized to the head and neck region

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Lingual Tonsil Size | 3 months
  Lingual tonsil tissue size will be measured on computed tomography image at baseline and remeasured following CT imaging after 3 months of proton pump inhibitor therapy.

SECONDARY OUTCOMES:
Calgary Sleep Apnea Quality of Life Index | 1, 2 and 3 months
  Calgary Sleep Apnea Quality of Life Index measures the quality of life in sleep apnea patients.
Visual Analog Scale of snoring | 1, 2 and 3 months
  Visual Analog Scale of snoring measures the loudness and disturbance factor related to snoring as documented by the bedpartner (when available)
Epworth Sleepiness scale | 1, 2 and 3 months
  Epworth Sleepiness scale measures the daytime sleepiness caused by sleep disturbances and interruptions associated with sleep apnea or snoring.
Reflux Symptom Index | 1, 2, and 3 months
  Reflux Symptom Index monitrors the physical signs and symptoms of laryngopharyngeal reflux during treatment obtained during fiberoptic endoscopy of the larynx, pharynx and esophagus.
Laryngopharyngeal Reflux | 3 months
  Continuous 24 hour laryngopharyngeal pH monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Michael Friedman, MD, Principal Investigator — Head and Neck and Cosmetic Surgery Inc and Advanced Center for Specialty Care; Ninos J Joseph, BS, Study Director — Advanced Center for Specialty Care
Locations (1):
- Advanced Center for Specialty Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Jamieson JR, Stein HJ, DeMeester TR, Bonavina L, Schwizer W, Hinder RA, Albertucci M. Ambulatory 24-h esophageal pH monitoring: normal values, optimal thresholds, specificity, sensitivity, and reproducibility. Am J Gastroenterol. 1992 Sep;87(9):1102-11. PMID 1519566
- [Background] DelGaudio JM, Naseri I, Wise JC. Proximal pharyngeal reflux correlates with increasing severity of lingual tonsil hypertrophy. Otolaryngol Head Neck Surg. 2008 Apr;138(4):473-8. doi: 10.1016/j.otohns.2007.12.023. PMID 18359357
- [Background] Mamede RC, De Mello-Filho FV, Vigario LC, Dantas RO. Effect of gastroesophageal reflux on hypertrophy of the base of the tongue. Otolaryngol Head Neck Surg. 2000 Apr;122(4):607-10. doi: 10.1067/mhn.2000.98362. PMID 10740190
- [Background] Dundar A, Ozunlu A, Sahan M, Ozgen F. Lingual tonsil hypertrophy producing obstructive sleep apnea. Laryngoscope. 1996 Sep;106(9 Pt 1):1167-9. doi: 10.1097/00005537-199609000-00022. PMID 8822724
- [Background] Suzuki K, Kawakatsu K, Hattori C, Hattori H, Nishimura Y, Yonekura A, Yagisawa M, Nishimura T. Application of lingual tonsillectomy to sleep apnea syndrome involving lingual tonsils. Acta Otolaryngol Suppl. 2003;(550):65-71. doi: 10.1080/0365523031000057. PMID 12737346
- [Background] Fricke BL, Donnelly LF, Shott SR, Kalra M, Poe SA, Chini BA, Amin RS. Comparison of lingual tonsil size as depicted on MR imaging between children with obstructive sleep apnea despite previous tonsillectomy and adenoidectomy and normal controls. Pediatr Radiol. 2006 Jun;36(6):518-23. doi: 10.1007/s00247-006-0149-7. Epub 2006 Apr 5. PMID 16596369
- [Background] Friedman M, Wilson MN, Pulver TM, Golbin D, Lee GP, Gorelick G, Joseph NJ. Measurements of adult lingual tonsil tissue in health and disease. Otolaryngol Head Neck Surg. 2010 Apr;142(4):520-5. doi: 10.1016/j.otohns.2009.12.036. PMID 20304271
- [Background] Wise SK, Wise JC, DelGaudio JM. Gastroesophageal reflux and laryngopharyngeal reflux in patients with sleep-disordered breathing. Otolaryngol Head Neck Surg. 2006 Aug;135(2):253-7. doi: 10.1016/j.otohns.2006.05.012. PMID 16890078
- [Background] Friedman M, Gurpinar B, Lin HC, Schalch P, Joseph NJ. Impact of treatment of gastroesophageal reflux on obstructive sleep apnea-hypopnea syndrome. Ann Otol Rhinol Laryngol. 2007 Nov;116(11):805-11. doi: 10.1177/000348940711601103. PMID 18074664
- [Background] Senior BA, Khan M, Schwimmer C, Rosenthal L, Benninger M. Gastroesophageal reflux and obstructive sleep apnea. Laryngoscope. 2001 Dec;111(12):2144-6. doi: 10.1097/00005537-200112000-00012. PMID 11802013
- [Background] Farrokhi F, Hill EM, Sun G, et al. Dx-pH Monitoring: how does it compare to the standard pH probe? Am J Gastroenterol 2007;103:S2.
- [Background] Reichel O, Dressel H, Wiederanders K, Issing WJ. Double-blind, placebo-controlled trial with esomeprazole for symptoms and signs associated with laryngopharyngeal reflux. Otolaryngol Head Neck Surg. 2008 Sep;139(3):414-20. doi: 10.1016/j.otohns.2008.06.003. PMID 18722223
- [Background] Park W, Hicks DM, Khandwala F, Richter JE, Abelson TI, Milstein C, Vaezi MF. Laryngopharyngeal reflux: prospective cohort study evaluating optimal dose of proton-pump inhibitor therapy and pretherapy predictors of response. Laryngoscope. 2005 Jul;115(7):1230-8. doi: 10.1097/01.MLG.0000163746.81766.45. PMID 15995512